CLINICAL TRIAL: NCT00626379
Title: Low CV Risk, Ages 25-44 & CV/Non-CV Outcomes, Ages 65+
Brief Title: Examining How Heart Disease Risk Factors Affect Healthy Aging (The Chicago Healthy Aging Study [CHAS])
Acronym: CHAS
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1379; R01HL081141-04 (NIH)
Record Dates: First submitted 2008-02-27; First posted 2008-02-29 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Coronary Disease; Cardiovascular Diseases
Keywords: Coronary Heart Disease; Subclinical Atherosclerosis; CVD-Related Markers of Inflammation; Mortality
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
Heart disease is the leading cause of death in the United States and is responsible for 30% of all deaths in the United States. This study will examine how risk factors for heart disease in young and middle aged people affect people's health as they grow older.

DETAILED DESCRIPTION:
Heart disease, including coronary heart disease (CHD) and cardiovascular disease (CVD), is a serious health problem in the United States. It is the leading cause of death in this country, and each year almost 700,000 people die from the disease. Risk factors for heart disease include high blood pressure, high cholesterol levels, tobacco use, diabetes, and history of a prior heart attack. It has been shown that young and middle aged adults with few risk factors experience a lower incidence of heart disease, lower Medicare costs, and longer lives than those with more risk factors. However, it is not known how having a low risk for heart disease at a young age affects health-related outcomes in older age. It may be possible that a low risk for developing heart disease in younger years results in healthier aging than does a higher risk. This study will examine former participants of the Chicago Heart Association (CHA) study who are now 65 to 84 years old. The purpose of this study is to determine how risk factors for heart disease in young adulthood and middle age are related to healthy aging.

This study will enroll 1500 people who participated in the CHA study from 1967 to 1973 and who are still living in the Greater Chicagoland area. Six hundred former participants who had a low risk of developing heart disease and 900 former participants who had a high risk of developing heart disease will be enrolled. Participants will attend one study visit that will include medical history interviews and questionnaires, a physical examination, blood pressure measurements, blood and urine collection, and an electrocardiogram (ECG) to measure the electrical activity of the heart. Blood samples will be collected and stored for future genetic testing. Participants will undergo physical functioning performance tests on balance, leg strength and coordination, grip strength, and endurance. They will also undergo a computed tomography chest scan to measure the amount of calcium in the arteries of the heart and ultrasound scans of the arteries in the neck to measure artery size and function.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the CHA study
* Lives in the Greater Chicagoland area

Exclusion Criteria:

* Severely ill, disabled, or cognitively impaired

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Original participants in the Chicago Heart Association (CHA) Detection in Industry study (1967 to 1973) who still reside in the Greater Chicagoland area.
Sampling Method: Probability Sample
Enrollment: 1395 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Subclinical atherosclerosis, CVD-related markers of inflammation, and levels of physical performance | Measured during participant's one (baseline) study visit

CONTACTS AND LOCATIONS:
Overall Officials: Martha L. Daviglus, MD, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Preventive Medicine Research Clinic, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share.